CLINICAL TRIAL: NCT02357758
Title: Recurrent Urinary Tract Infections in Children: Bacterial Identification, Antibiotic Susceptibility Profiling and Cytokine Levels Associated With Antibiotic Prophylaxis
Brief Title: Effects of Antibiotic Prophylaxis on Recurrent UTI in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R-12-387
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2015-09

CONDITIONS: Urinary Tract Infection; Recurrent Urinary Tract Infection
Keywords: Antibiotic Prophylaxis; Urinary Microbiota
MeSH Terms: conditions — Urinary Tract Infections | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Antibiotic Prophylaxis (Active Comparator): Patients with RUTI receiving Septra (Trimethoprim dose 2mg/kg) or nitrofurantoin (dose 2 mg/kg) as determined by clinician.
  Interventions: Drug: Antibiotic Prophylaxis
- Healthy Population (No Intervention): Healthy population
- Clinical Observation (No Intervention): Patients experiencing RUTI that do not require antibiotic prophylaxis as determined by clinician.

INTERVENTIONS:
Drug: Antibiotic Prophylaxis — Approved clinical dosage or antibiotics
  Arms: Antibiotic Prophylaxis

SUMMARY:
Approximately, 3% of males and 8% of females will develop a urinary tract infection (UTI) during childhood, and most of these will be effectively treated by short-term antibiotic therapy. A subset of these children (20-48%), will develop recurrent UTI (RUTI), which may have long-term effects in the form of hypertension or renal damage.

In an effort to prevent RUTIs physicians prescribe sulfamethoxazole-trimethoprim (Septra) or nitrofurantoin as low dose antibiotic prophylaxis. However, recent evidence suggests that during prophylactic therapy the body is exposed to antibiotic levels capable of increasing antibiotic resistance and bacterial virulence. This has been shown to be true in the uropathogens E. coli and Staphylococcus saprophyticus, yet it is not known if Enterococcus sp. demonstrate similar mechanisms. Additionally, antibiotics have been shown to disrupt the natural balance of the human microbiome, potentially leading to major long term problems.

As a uropathogen, enterococci consistently rank in the top 3 causes of RUTI, especially in children under 3 years of age. Additionally, Enterococcus is notorious for developing antibiotic resistance and studies have shown that children with enterococcal UTIs exhibit a higher rate of recurrence than those with non-enterococcal UTIs.

The investigators hypothesize the current practice of antibiotic prophylaxis in children with RUTI is detrimental and can change the bacterial and sensitivity profiles of these patients.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria will be recruited to the study at Dr. Dave's discretion through the urology clinic. As clinically indicated patients will then fall into one of two groups, patients receiving antibiotic prophylaxis or those undergoing clinical observation. This reflects the standard of care these children receive and no additional procedures are mandated.

At the initial appointment information sheets and consent forms will be given to the parent/caregiver to consider; due to the nature of the study, the parent or legal guardian will be required to give informed consent. Following the receipt of informed consent, patients will be asked to provide a mid stream urine sample given they are infection free and not currently on antibiotics. Patients will be assessed simultaneously for dysfunctional elimination syndrome (DES) through review of their 48-hour bowel bladder diary, the completed Dysfunctional Voiding Scoring System (DVSS) questionnaire and performing uroflowmetry. Patients may withdraw from the study at any stage without repercussion.

Patients in the antibiotic prophylaxis group will receive a 3-month script for antibiotic prophylaxis, if clinically indicated according to the standard of care. Septra (Trimethoprim dose 2 mg/kg) or nitrofurantoin (dose 2 mg/kg) will be the antibiotics used for prophylaxis based on past cultures or allergy history. Antibiotic prescription will be renewed at 3 months and an informal assessment on compliance will be performed through review of the number of doses left. Patients not tolerating one of these antibiotics will be offered the alternate. From months 6-12, prophylaxis will cease (washout period) unless a symptomatic UTI is suspected at which point appropriate treatment will be implemented. Lifestyle changes, behavioural modification and management of constipation will be instituted in both groups. Patients will return for follow up visits at 3, 6, 9 and 12 months. In addition, patients can return to the urology clinic at any time if UTI is suspected.

Urine samples will be collected at baseline and at 3, 6, 9 and 12 months from both groups (prophylaxis versus observation) by registered nurses at Children's Hospital, London Health Sciences Centre. Healthy patients, those with no recent history of UTI or antibiotic use or known urinary tract abnormalities, will be included to give an indication of the healthy urinary microbiota in the paediatric population. These participants will be asked to provide urine at two time points a minimum of three months apart. Samples will be assessed for bacterial identification via both culture dependent and independent methods. Antibiotic susceptibility profiles will be determined for viable organisms using the Kirby Bauer disk method and bacterial virulence analyzed via bladder and kidney cell line adherence and internalization assays, as well as PCR to determine the presence of virulence genes associated with the pathogen (adhesins, fimbriae, toxins). Urinary cytokine analysis via Luminex will also be conducted as a measure of host bladder state, immune response and disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Patient has experienced a minimum of 2 UTIs within the last year, as well as a culture proven UTI for inclusion into either of the RUTI groups.
* Patients must be deemed to require antibiotic prophylaxis, at the discretion of Dr. Dave and following the standard of care, for inclusion in the antibiotic prophylaxis group.
* Patients with no known urological abnormalities, recent history of UTI or antibiotic use are eligible for inclusion in the healthy patient group.

Exclusion Criteria:

* Patients with an abnormal urinary tract as determined through the use of ultrasound and, given an abnormal ultrasound, or greater than two febrile UTIs, a voiding cystourethrogram (VCUG). The use of both ultrasound and VCUG given these indications is standard of care.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Dave, MD, MCh, Principal Investigator — Assistant Professor, Pediatric Urologist, London Health Sciences Centre
Locations (1):
- Children's Hospital - London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Whiteside SA, Dave S, Seney SL, Wang P, Reid G, Burton JP. Enterococcus faecalis persistence in pediatric patients treated with antibiotic prophylaxis for recurrent urinary tract infections. Future Microbiol. 2018 Aug;13:1095-1115. doi: 10.2217/fmb-2018-0048. Epub 2018 Aug 22. PMID 30132694

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiotic Prophylaxis: Patients with RUTI receiving Septra (Trimethoprim dose 2mg/kg) or nitrofurantoin (dose 2 mg/kg) as determined by clinician.
  Antibiotic Prophylaxis
Period: Overall Study
Arm/Group | Antibiotic Prophylaxis | Healthy Population | Clinical Observation
Started | 25 | 20 | 12
Completed | 9 | 20 | 5
Not Completed | 16 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotic Prophylaxis | Healthy Population | Clinical Observation | Total
Number analyzed (Participants) | 25 | 20 | 12 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 20 | 12 | 57
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 12 | 57
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 20 | 12 | 57

OUTCOME MEASURES:

1. Primary Outcome: Changes to the Urinary Microbiota
Description: Changes to the urinary microbiota were measured as changes in the colony forming units (CFUs) of Enterococcus sp., Escherichia coli, Klebsiella sp./Enterobacter sp., Staphylococcus saprophyticus, or Pseudomonas sp./Staphylococcus aureus when the participant urine was cultured on CHROMagar Orientation. The data was analyzed in terms of bacterial counts, presence/absence, and presence at or above the diagnostic threshold for UTI (10^5 CFU/mL of one species). Here we present participant midstream urine samples that met the diagnostic threshold for UTI at baseline.
Time Frame: Baseline, 3-, 6-, 9-, 12-months
Population: Bacterial culture data was not available for all participants due to the low volume of some samples.
Measure: Number; unit: participants
Groups:
- Healthy Population: Patients with no history of RUTI or recent antibiotic usage.
Arm/Group | Antibiotic Prophylaxis | Healthy Population | Clinical Observation
Number analyzed (Participants) | 17 | 19 | 10
participants | 3 | 2 | 1

2. Secondary Outcome: Changes to Metabolic Profiles of Urine
Description: Changes to metabolic profiles of urine as determined using gas chromatography mass spectrometry (GC-MS).
Time Frame: Baseline, 3-, 6-, 9- 12-months
Reporting Status: Not Posted

3. Secondary Outcome: Changes to Antibiotic Susceptibility
Description: Changes to antibiotic susceptibility of cultured bacteria as determined by the Kirby Bauer disc diffusion method.
Time Frame: Baseline, 3-, 6-, 9-, 12-months
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Pro-inflammatory Cytokines
Description: Changes in pro-inflammatory cytokines associated with inflammation and immune cell recruitment will be measured using multiplexed immunoassay kits employing Luminex® xMAP fluorescent beadbased technology.
Time Frame: Baseline, 3-, 6-, 9-, 12-months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year - Over the course of prophylaxis or clinical observation.
Description: Adverse events were reported according to the clinicaltrials.gov definitions.
  Adverse event information was collected during clinical appointments.
Arm/Group | Antibiotic Prophylaxis | Healthy Population | Clinical Observation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/19 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/19 | 0/12
Other Adverse Events (participants affected / at risk) | 0/25 | 0/19 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No